CLINICAL TRIAL: NCT03327506
Title: Efficacity of Hypnosis Versus Premedication for the Management of Perioperative Anxiety in Gynecological Surgery
Brief Title: Preoperative Hypnosis Versus Premedication in Gynecological Surgery
Acronym: HYPNOGYN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-002112-13
Record Dates: First submitted 2017-10-17; First posted 2017-10-31 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Gynecologic Disease; Anxiety Disease
Keywords: Premedication/ Hypnosis/ Anxiety/Surgery
MeSH Terms: conditions — Genital Diseases, Female | interventions — Alprazolam; Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypnosis group (Experimental): Intervention: hypnosis session the eve of the surgery
  Interventions: Drug: Alprazolam 0.5 mg
- premedication (Active Comparator): alprazolam 0,5 mg the eve and the morning of the surgery
  Interventions: Drug: Alprazolam 0.5 mg

INTERVENTIONS:
Drug: Alprazolam 0.5 mg — alprazolam 0,5 mg the eve and the morning of the surgery versus a preoperative hypnosis session
  Other Names: hypnosis

SUMMARY:
The aim of this study is to evaluate the efficacy of an hypnosis session, performed on the eve of a laparoscopic gynecological surgery, on the level of immediate preoperative anxiety measured by State-Trait Anxiety Index (STAI-Y) self-administered questionnaire compared to premedication by alprazolam®.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age: over 18 years
* Patient care and follow-up at the regional maternity center of Nancy (CHRU of Nancy)
* Female patient for whom gynecological laparoscopic surgery is programmed and lasting longer than 1 hour (ovarian cyst, laparoscopy infertility, laparoscopic promontofixation, noncarcinogenic assisted laparoscopy hysterectomy, endometriosis, diagnostic laparoscopy, pyosalpinx, hydrosalpinx)
* Patient with Physical status score (ASA) score between 1 and 3
* With standardized anesthesia protocol
* Patient affiliated to a Social Security
* Patient has received complete information about the organization of the research and has signed her informed consent

Exclusion Criteria:

* Pretreatment by benzodiazepines
* Known hypersensitivity to Alprazolam® (including undocumented)
* Prohibition conditions to Alprazolam®: Severe respiratory insufficiency, Sleep apnea syndrome, Myasthenia, Severe acute or chronic hepatic impairment
* Ongoing major depressive episode
* Chronic use (> 1 month) of benzodiazepines or morphine or analgesics of level 2
* Participation in a therapeutic trial 6 months before inclusion in this trial
* Patient referred to in Articles L. 1121-5 to L. 1121-8 and L1122-2 of the Public Health Code

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Preoperative Anxiety score evaluated by STAI-Y | before surgery (day 2_before)
  evaluated by STAI-Y self-administered questionary

SECONDARY OUTCOMES:
Anxiety score evaluated by analogue visual scale | at inclusion visit (day 1), before surgery (day 2_before), after surgery (day 2_after), 24 h after the surgery (day 3)
  evaluated by analogue visual scale (EVA 0 to 10)
sleep quality evaluated by EVA scale | day 2_before and the day 3
  evaluated by EVA scale (0 to 10)
patient satisfaction score evaluated by EVA scale | day 3
  evaluated by EVA scale (0 to 10)
analysis of salivary amylase | day 1 and day2_before
  salivary amylase
postoperative fatigue evaluated by EVA scale | day 3
  evaluated by EVA scale (0 to 10)
Intraoperative morphine and hypnotics drugs Consumption | day 3
  Consumption
Incidence of nausea and vomiting | day 3
  Incidence
Score of pain measured by EVA scale | day 2_after, day 2_recovery room (at the end of recovery room) and Day 3
  measured by EVA (0 to 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Florence Vial, Nancy, France